CLINICAL TRIAL: NCT00913211
Title: rTMS and Motor Learning Training to Promote Recovery From Hemiparesis
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) to Promote Hand Recovery in Stroke
Acronym: rTMS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0704M06701; 1R01HD053153-01A2 (NIH)
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- rTMS only (Experimental): brain stimulation to non-stroke primary motor area
  Interventions: Device: rTMS
- Finger tracking training (Experimental): Motor learning training using finger flexion/extension tracking movements toward a target.
  Interventions: Procedure: Motor learning training
- rTMS and finger tracking (Experimental): Combination of rTMS and tracking
  Interventions: Procedure: rTMS and Tracking
- Sham (Placebo Comparator): Sham rTMS treatment
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: rTMS — 600 pulses of 6 hz priming rTMS at 90% of threshold followed by 600 pulses of low-frequency rTMS at 90% of threshold.
  Arms: rTMS only
Procedure: Motor learning training — one hour of repeated finger tracking movements toward a changing target.
  Arms: Finger tracking training
Procedure: rTMS and Tracking — Combination of rTMS and finger tracking
  Arms: rTMS and finger tracking
Device: Sham rTMS — Sham treatment of rTMS
  Arms: Sham

SUMMARY:
Paralysis following stroke stems not only from the loss of neurons killed by the stroke but also from the loss of neurons lying dormant in the stroke hemisphere. One of the reasons viable neurons become dormant (down-regulated) is because of excessive interhemispheric inhibition imposed on them from the nonstroke hemisphere. The challenge in neurorehabilitation is to restore excitability and voluntary control of these down-regulated neurons in the stroke hemisphere. Suppression of the source of this excessive interhemispheric inhibition can be achieved with the noninvasive method called repetitive transcranial magnetic stimulation (rTMS). It has been shown in healthy subjects that the known depressant effects of low-frequency rTMS can be increased and prolonged by preceding it with 6-Hz priming stimulation. In a recent safety study, we showed that one treatment of 6-Hz primed low-frequency rTMS applied to the nonstroke hemisphere is safe. It is now important to evaluate a series of these treatments and whether their efficacy can be enhanced by combining the rTMS with motor learning training. The specific aims of this study are to determine the efficacy, mechanism, and safety of a series of 5 treatments of 6-Hz primed low-frequency rTMS applied to nonstroke hemisphere and combined with motor learning training to promote recovery of the paretic hand. Forty subjects with stroke will be randomly assigned to one of four treatment groups. The rTMS/only group will receive 20 min. of rTMS per day. The Track/only group will receive 20 min. of finger tracking training per day. The rTMS/combined group will receive alternating days of the rTMS and Track treatments. The rTMS/sham group will receive 20 min. of rTMS using a sham electrode each day. The hypotheses are: 1) the rTMS/combined group will show the greatest improvements in hand function, 2) the rTMS/combined group will show the greatest improvements in cortical excitability using paired-pulse TMS testing and in brain reorganization using fMRI, and 3) the rTMS treatment will be safe. The proposed research is important because it addresses the greatest cause of long-term disability in society, hemiparesis following stroke, and it is innovative because it applies a technique never used before, 6-Hz primed low-frequency rTMS combined with motor learning training. The potential impact of this research is a radical change to rehabilitation that accomplishes a higher quality of life in stroke.

DETAILED DESCRIPTION:
The proposed research penetrates the problem of hemiparesis following stroke. This problem devastates quality of life in thousands of people each year. The brain shows remarkable ability to reorganize under certain conditions, including after stroke. Unfortunately, some changes are maladaptive and leave the individual with additional loss of function beyond that caused directly by the ischemic damage. Specifically, motor neurons in the ipsilesional (stroke) hemisphere that have survived the stroke can undergo a loss of excitability due to exaggerated interhemispheric inhibition imposed on them from neurons in the contralesional (non-stroke) hemisphere through transcallosal pathways. Fortunately, the maladaptive reorganization is reversible, even in chronic stroke, through forced-use and forced-learning paradigms with the paretic limb. But we postulate that the effectiveness of behavioral training can be richly enhanced when combined with electrophysiologic intervention that also affects neural excitability. Repetitive transcranial magnetic stimulation (rTMS) is a potent and noninvasive way to influence the excitability of the brain. rTMS, at low stimulation frequencies, depresses neural function. By stimulating the contralesional motor cortex at low frequency, thereby depressing interhemispheric inhibition, a net excitatory effect (disinhibition) is induced upon the ipsilesional motor cortex. Furthermore, it has been shown in animals and in healthy humans that the depressive effect on the stimulated hemisphere can be magnified by preceding the low-frequency rTMS with 6-hz "priming" rTMS. We will call this arrangement 6-Hz primed low-frequency rTMS. We contend that by combining 6-Hz primed low-frequency rTMS with behavioral motor learning training unprecedented improvements in recovery from hemiparesis can be achieved. We have recently demonstrated the safety of a single treatment of 6-Hz primed low-frequency rTMS in stroke but a large gap in knowledge still exists in not knowing the effect of serial treatments of 6-Hz primed low-frequency rTMS combined with motor learning training. Failure to address this gap only perpetuates the use of conservative strategies in stroke rehabilitation, which may rob individuals of their fullest possible recovery.

Our long-term goal is to maximize motor recovery following stroke. The objective of this proposal is to integrate the excitability effects induced exogenously by rTMS with those produced endogenously by motor learning to produce a powerful yet safe interactive effect leading to improved recovery from hemiparesis. The central hypothesis is that serial treatments of 6-Hz primed low-frequency rTMS combined with motor learning training will be effective and safe. Our research team is uniquely qualified to execute this project because of 1) special training in rTMS undertaken by the PI in the laboratory of an international leader in rTMS, 2) participation of this leader as a consultant, 3) participation of a neuroscientist with expertise in stroke neuroplasticity as a consultant, 4) participation of a recognized expert in cerebrovascular disease as a co-investigator, 5) conducting the study in the University of Minnesota's General Clinical Research Center to maximize protection of patients, and 6) inclusion of the Center for Magnetic Resonance Research for studying brain reorganization.

The specific aims of this project are to:

Specific Aim #1. Determine the efficacy of using serial treatments of 6-Hz primed low-frequency rTMS, in isolation and in combination with motor learning training, to improve hand function in stroke.

Forty subjects with stroke (with partial movement in weak hand, able to walk 100 feet, able to follow directions, no history of seizures, no medical devices or metal incompatible with mri) will be randomly assigned in equal numbers to one of four treatment groups: The rTMSonly group will receive 5 treatments of rTMS to the primary motor area (M1) of the contralesional hemisphere consisting of 10 min. of 6-Hz ("priming") rTMS at 90% of resting motor threshold interrupted into 20 trains of 5-s duration with 25-s intervals between trains then followed immediately by 10 additional min. of 1-Hz ("low-frequency") rTMS continuously at 90% of resting motor threshold. Treatments will be every other day over two weeks. The Trackonly group will receive 5 treatments of computerized finger tracking training every other day for two weeks. The rTMScombined group will receive the same rTMS as the rTMSonly group and it will be alternated with the same tracking training as the Trackonly group until 5 days of each have occurred over a two-week period. The rTMSsham group will receive the same rTMS procedures, including similar sound, but no magnetic stimulation will occur. The four treatments have a 2x2 factorial design, with rTMS and tracking as the factors, which allows estimation of any synergistic effects of rTMS combined with tracking. Behavioral gains in the paretic hand will be measured with finger prehension/dexterity tests, finger tracking accuracy, subject self ratings and examiner ratings. The working hypotheses are:

1. the rTMScombined group will show greater improvements in paretic hand function than the rTMSonly and Trackonly groups at posttest and at one-month follow-up, and
2. the rTMSonly and Trackonly groups will show greater improvements than the rTMSsham group.

Specific Aim #2. Explore the neural mechanism associated with 6-Hz primed low-frequency rTMS combined with tracking training.

Following the treatments described in Aim #1, M1 excitability will be measured with paired-pulse TMS testing in the ipsilesional hemisphere. This testing will allow for examination of both cortical inhibition and excitation. In addition, brain reorganization associated with voluntary activation will be measured with functional MRI yielding data on volume and signal intensity of active voxels during paretic finger tracking. The working hypotheses are:

1. the rTMScombined group will show greater increases in cortical excitability and brain reorganization in the ipsilesional hemisphere than the rTMSonly and Trackonly groups at posttest and at one-month follow-up,
2. the rTMSonly and Trackonly groups will show greater increases than the rTMSsham group.

Specific Aim #3. Determine the safety of serial 6-Hz primed low-frequency rTMS treatments in stroke.

Associated with the treatments described in Aim #1, adverse effects will be measured through observation for seizures at the time of treatment. Neurocognitive tests will measure mood, verbal comprehension, perceptual organization, working memory and processing speed. Also, a finger tracking test will measure motor control in the nonparetic hand. The working hypothesis is:

1. five 6-Hz primed low-frequency rTMS treatments, given alone or in combination with motor learning training, will not produce any seizure activity or any other serious adverse effect.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke at least 6 months prior, partial movement of paretic hand, ability to follow directions, ability to walk 100 feet, motor evoked response in stroke hemisphere during TMS

Exclusion Criteria:

* No history of seizures, no medical devices or metal incompatible with fMRI

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
box and block finger prehension test | 45 days

SECONDARY OUTCOMES:
cortical excitability | from pretest to posttest (2 weeks)
  Paired pulse TMS testing will show increase in the ratio of paired pulse to single pulse MEP amplitude when stimulating ipsilesional M1.
cognitive function | pretest to posttest (2 weeks)
  There will be no decline in function on the Hopkins Verbal learning test.

CONTACTS AND LOCATIONS:
Overall Officials: James R Carey, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States